CLINICAL TRIAL: NCT04804748
Title: Safety and Efficacy of Low-energy Electrical Cardioversion With or Without Bi-atrial Pacing in Patients With Post-operative Atrial Fibrillation in a Real World Setting - The DefiPace Study
Brief Title: The DefiPace Study
Acronym: Defipace
Status: Recruiting | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Collaborators: Osypka AG (Unknown)
Responsible Party: Sponsor
Other Study IDs: IPPMed Defipace 202103
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Post-operative Atrial Fibrillation POAF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase A: Approximately 150 consecutive patients undergoing elective cardiac surgery (bypass and / or valve surgery)
  * Data regarding standard of care post-operative pacing and treatment of POAF, if applicable, will be collected from time of surgery until discharge
  * No use of an external bi-atrial pacing device
  * No use of Defipace
  * In-hospital data will be collected for all patients
  * Patients that developed POAF (n=50) will be followed-up with a phone call 30 days after surgery
  Interventions: Other: No intervention
- Phase B: Approximately 300 consecutive patients undergoing elective cardiac surgery (bypass and / or valve surgery) with planned TMA implantation
  * In-hospital data will be collected for all patients
  * Use of the DefiPace system for the treatment (low-energy cardioversion) and post-operative prevention (bi-atrial pacing) of POAF will be documented (n=100). These patients will be followed-up with a phone call 30 days after surgery
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no intervention

SUMMARY:
Prospective, non-interventional, multi-center, international registry in two phases in consecutive patients undergoing elective cardiac surgery.

The DefiPace registry is designed in two phases

1. to document the standard of care in 50 patients with atrial fibrillation (AF)
2. to assess the treatment and outcomes of patients with post-operative atrial fibrilllation using low-energy cardioversion and subsequent bi-atrial pacing in clinical practice in 100 patients

DETAILED DESCRIPTION:
Phase A Approximately 150 consecutive patients undergoing elective cardiac surgery (bypass and / or valve surgery)

* Data regarding standard of care post-operative pacing and treatment of POAF, if applicable, will be collected from time of surgery until discharge
* No use of an external bi-atrial pacing device
* No use of Defipace
* In-hospital data will be collected for all patients
* Patients that developed POAF (n=50) will be followed-up with a phone call 30 days after surgery.

Phase B Approximately 300 consecutive patients undergoing elective cardiac surgery (bypass and / or valve surgery) with planned TMA implantation

* In-hospital data will be collected for all patients
* Use of the DefiPace system for the treatment (low-energy cardioversion) and post-operative prevention (bi-atrial pacing) of POAF will be documented (n=100). These patients will be followed-up with a phone call 30 days after surgery

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled to undergo elective open chest cardiac surgery (bypass and / or valve surgery)
* Patient is at least 18 years old
* Patient with isolated bypass surgery is at least 70 years old
* Patient with valve surgery is at least 60 years old
* Patient provides written informed consent prior to the procedure
* Phase B only: patient is scheduled for TMA implantation during the elective cardiac surgery and is potentially eligible for DefiPace use

Exclusion Criteria:

* Clinical history of either permanent, persistend or paroxysmal atrial fibrillation
* Permanent pacemaker/defibrillator, other intra-cardiac active implanted electronic devices
* Minimally-invasive surgery
* Recent stroke within the last 3 months
* A history of or current endocarditis
* Pregnacy at the time of surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Phase A Approximately 150 consecutive patients undergoing elective cardiac surgery (bypass and / or valve surgery) Phase B Approximately 300 consecutive patients undergoing elective cardiac surgery (bypass and / or valve surgery) with planned TMA implantation.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of POAF | 30 days
  Incidence of POAF
Termination of POAF | 30 days
  Termination of POAF
Time in POAF | 30 days
  Time in POAF (AF Burden)
Time to cardioversion | 30 days
  Median time to cardioversion
Number of shocks | 30 days
  Mean number of shocks per patient
Energy requirements | 30 days
  Mean energy requirements (first/subsequent)
POAF recurrence | 30 days
  POAF recurrence/repeat cardioversions
Time in ICU | 30 days
  Time in ICU in hours
Procedural success | 30 days
  Procedural success
Time needed for electrode placement | 30 days
  Time needed for electrode placement

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bramlage, Professor, Study Director — IPPMed
Locations (10):
- Medical University of Vienna, Vienna, Austria
- Germany (9):
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Klinikum Nürnberg, Nuremberg, Bavaria
  - University Hospital of Würzburg, Würzburg, Bavaria
  - Oldenburg Hospital AöR / Medical Campus University of Oldenburg, Oldenburg, Lower Saxony
  - Heart Center Dresden GmbH University Hospital, Dresden, Saxony
  - Albert-Ludwigs-Universitaet Freiburg, Freiburg im Breisgau
  - Hannover Medical School, Hanover
  - University Hospital Jena, Jena
  - University Hospital Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bechtel JF, Christiansen JF, Sievers HH, Bartels C. Low-energy cardioversion versus medical treatment for the termination of atrial fibrillation after CABG. Ann Thorac Surg. 2003 Apr;75(4):1185-8. doi: 10.1016/s0003-4975(02)04715-x. PMID 12683560
- [Background] Liebold A, Wahba A, Birnbaum DE. Low-energy cardioversion with epicardial wire electrodes: new treatment of atrial fibrillation after open heart surgery. Circulation. 1998 Sep 1;98(9):883-6. doi: 10.1161/01.cir.98.9.883. PMID 9738643